CLINICAL TRIAL: NCT06419387
Title: The Effect of Flash Technique Via Self-Therapy App on Depression, Anxiety, and Traumatic Symptoms in Individuals Who Have Experienced a Traffic Accident: A Randomized-Controlled Design
Brief Title: The Effect of Flash Technique Via Self-Therapy App on Depression, Anxiety, and Traumatic Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Therapeutic Sciences, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBA2024
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Stress Disorder
Keywords: EMDR; Mobile App; Traumatic Stress
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: EMDR Mobile App (Intervention) Group vs. Psycho-educational (Video) Control Group
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Therapy App (Experimental): EMDR Flash Technique protocol will be administered via Self-Therapy App.
  Interventions: Device: Self-Therapy Mobile App
- Psycho-Education (Active Comparator): Psycho-Education will be administered via videos of a psychology professor.
  Interventions: Other: Psycho-education Videos

INTERVENTIONS:
Device: Self-Therapy Mobile App — Self-Therapy Mobile App includes videos and guidelines for applying EMDR Flash Technique
  Arms: Self-Therapy App
Other: Psycho-education Videos — Psycho-education Videos include guidelines for increasing emotion regulation skills.
  Arms: Psycho-Education

SUMMARY:
EMDR is a psychotherapy method utilized for treating psychological traumas, with the Flash technique being one of its quickest and most effective methods. The "Self-Therapy" mobile application, accessible via Apple Store and Google Play, enables users to self-administer the Flash technique, following specific guidelines to help reduce symptoms like depression, anxiety, and stress linked to traumatic memories. Designed for adults over 18, particularly those diagnosed with mental health disorders, it is advised to be used under a psychiatrist's guidance. The application features a virtual guide, an avatar named Therapist Yağmur, who assists users through the process, including relaxation exercises and progress tracking. This allows users to pause and resume therapy as needed. Such applications represent a significant advancement in remote psychological support, potentially increasing access to psychotherapy and fostering societal acceptance of psychological health services.

DETAILED DESCRIPTION:
EMDR is a psychotherapy method used in the treatment of psychological traumas. The Flash technique is considered one of the fastest and most effective techniques of EMDR. The self-therapy application allows users to apply the Flash technique by themselves by following guidelines, aiming to reduce depression, anxiety, and stress levels associated with traumatic memories. Applications like "Self-Therapy" could serve as an important model for the development and widespread adoption of remote psychological support services. With this project, individuals experiencing stressful life events could support their own healing process through a mobile application. This could lay the foundation for the development and expansion of similar mobile applications, thereby inspiring new projects and studies aimed at enhancing and increasing the accessibility of post-traumatic support services. The ease of access to psychotherapy through a mobile application could help increase societal awareness and acceptance of psychological health services.The "Self-Therapy" project is specifically designed for adults aged 18 and older who have experienced a traumatic or stressful event and perceive a decline in their quality of life due to its effects. The mobile application, available for download on both the Apple Store and Google Play, is primarily intended for individuals diagnosed with a mental health disorder, and it is recommended that they use the application under the guidance and recommendation of their psychiatrist.

The application employs a virtual guide, an avatar named Therapist Yağmur, who leads users through the program. Through the avatar's instructions, users engage in the Flash technique to actively address and work through their traumatic memories. Additionally, the application includes relaxation exercises that can be utilized as needed. Users are able to track their progress within the app, enabling them to pause and resume their therapeutic journey as required, thereby facilitating a self-directed approach to managing and potentially mitigating the impacts of their traumatic experiences.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Having access to the internet

Exclusion Criteria:

* A diagnosis of psychotic illness

  * Presence of mental retardation
* Moderate or severe depression
* Active suicidal thoughts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | 1-week and 1-month follow-up
  Depression, stress and anxiety scores will significantly change. Scores for depression, anxiety and stress are calculated by summing the scores. The scores are between 0-3, and more scores mean worse results.
  for the relevant items
Impact of Events Scale Revised (IES-R) | 1-week and 1-month follow-up
  Intrusion and hyperarousal scores will significantly change. The maximum mean score on each of the three subscales is '4', therefore the maximum 'total mean' IES- R score is 12. Lower scores are better.

CONTACTS AND LOCATIONS:
Locations (1):
- Academy of Therapeutic Sciences, Istanbul, Turkey (Türkiye)